CLINICAL TRIAL: NCT04907916
Title: The NAD Dependent Deacetylase Activity of Sirtuin1 in COVID19 Patients
Brief Title: Sirtuin1 in COVID19 Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, HHMHamed, Principal investigator, Assiut University
Other Study IDs: SIRTUIN1 in COVID19
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: SIRTUIN1 — The NAD dependent deacetylase activity of Sirtuin1

SUMMARY:
1. Evaluate serum level of NAD,Sirtuin1,ADAM17 andPARP1 in covid19 patients
2. Investigate the correlation between measured biomarkers and each other
3. Investigate the correlation between measured biomarkers and each other and their correlation with covid19 severity and outcome which may help in the therapy and prevention of disease complication(cytokine storm)

DETAILED DESCRIPTION:
December 2019, a number of cases of pneumonia with fever, cough, and dyspnea as clinical manifestations have been found in Wuhan, Hubei Province, China (Huang C et al., 2020) The analysis of the whole genome sequence of the respiratory samples suggests that it is a new type of betacoronavirus (Lu R, Zhao X, Li J et al ., 2020), which resembled severe acute respiratory syndrome coronavirus (SARS-CoV)] (Zhu N, Zhang D, Wang W et al .,2020). On February 11, 2020, the World Health Organization (WHO) officially named it coronavirus disease (COVID-19). COVID-19 may be asymptomatic or manifest in 3 clinical phases, an initial upper respiratory tract infection, with a few patients thereafter progressing to a pneumonic phase, and an even smaller number to the hyperinflammatory phase which may be lethal [ (Siddiqi H.K et al.,2020). The aim of any therapy would be to intervene at an early stage, either prophylactically or therapeutically, to prevent progression of the disease to a point where mechanical ventilation (MV) is required, or significant organ dysfunction occurs (Richards G et al., 2020).

Risk factors for a poor outcome include older age, comorbidity (in particular diabetes, hypertension and cardiac disease), non-asthmatic respiratory disease, obesity, immunosuppression and male sex (Williamson et al., 2020). The independent associations of advancing age, male sex, chronic respiratory conditions (though not well controlled asthma), chronic cardiac and chronic neurological disease with in-hospital mortality, are in line with other international reports - It is difficult however to determine why these conditions specifically are linked to mortality .(Clohisey S et al., 2019).

While the general concept of an excessive or uncontrolled release of pro-inflammatory cytokines is well known, an actual definition of what a hyperinflammatory response or "Cytokine Storm" In this phase, there is an unbalanced and exacerbated inflammatory response with the release of tumor necrosis factor (TNF-α), interleukin 1β (IL-1β), interleukin 6 (IL-6), as pro-inflammatory mediators together with interleukin 10 (IL-10) and interferon β as anti-inflammatory mediators. The complex interactions between TNF-α, the interleukins, chemokines and interferons in SARS-CoV-2 are currently poorly understood; however, they are associated with and related to a significant viraemia (Schultz M.B et al., 2016).

February 13, the journal ofRadiology has published several articles on the imaging features of COVID-19 (Chung M, Bernheim et al., 2019) but all of them are descriptive analyses. In February 2020, the Chinese Society of Radiology issued the radiologic diagnosis of pneumonia with COVID-19. CT plays an important role in the screening and diagnosis of COVID-19. The first edition of the experts (Lei J, Li J, Li X, Qi X et al., 2020)divided CT manifestations into three stages: early, progressive, and severe according to the extent and features of the pulmonary abnormalities. However, it did not clarify the relationship between the extent of inflammation and the clinical presentation of the patient. cases were divided into four groups: minimal, common, severe, and critical according to whether there were clinical symptoms, severity of pneumonia, respiratory failure, shock, other organ failure, etc., based on the Diagnosis and Treatment Plan of COVID-19 issued by National Health Commission (7th ed.) (in Chinese) (Fang Y, Zhang H et al., 2019). (1) Mild type: mild clinical symptoms without pneumonia in imaging; (2) common type: fever, respiratory tract and other symptoms with pneumonia in imaging; (3) severe type: respiratory distress, respiratory rate ≥ 30 times/min; in resting state, oxygen saturation ≤ 93%; NAD+ is a cofactor found in every cell of the body, and it is involved in multiple metabolic pathways. It is a fundamental housekeeping molecule that catalyses electron transfer in metabolic reduction-oxidation reactions, functioning as an electron shuttle in the production of adenosine triphosphate (ATP).

Sirtuins are an ancient family of seven NAD+-dependent deacylase and mono-ADP-ribosyl transferase signalling proteins that are intrinsically involved in metabolic regulation and cellular homeostasis. Of particular interest is SIRT1, which downregulates ADAM 17 (A Disintegrin and Metalloproteinase Domain 17), also called TNF-α converting enzyme (TACE), by increasing expression of TIMP3 the gene that encodes for tissue metalloproteinase inhibitor 3 [] (Fontani F et al., 2017) . In so doing it decreases levels of TNF-α, IL-1b and IL-6. An increase in TNF-α causes SIRT1 to down-regulate ADAM 17, thereby controlling TNF-α formation in a negative feedback loop that secondarily influences IL-1b and IL-6 production, which are dependent on TNF-α []. ADAM17 is a proteinase encoding gene. TNF-α and the cytokine receptor for IL-6 must be proteolytically cleaved in order to be systemically active, and ADAM17 provides this function. If ADAM17 expression is not downregulated by SIRT1, TNF-α and IL-6 are released, resulting in an uncontrolled hyperinflammatory response as may occur with COVID-19 (Cardellini M et al., 2009). SIRT 1, by inhibition of ADAM17 and thereby TNF-α and IL-6, performs an anti-inflammatory function . Upregulation of SIRT1 (Shin M.R et al., 2015) directly decreases viral replication and inhibits the activation of ADAM17, thereby decreasing TNF-α, IL-1b and IL-6. Conversely depletion of SIRT1 allows for increased viral replication with little or no inhibition of ADAM17 activity, causing uncontrolled increases in TNF-α, IL-6 and IL-1b. Whereas an increase in TNF-α would usually increase SIRT1 activity to downregulate ADAM17, in the presence of a deficiency of NAD+ or Zn++, this would not occur due to insufficient activation of SIRT1, causing an unchecked increase in TNF-α.

Increased age is a strong predictor of SARS-CoV-2-associated in-hospital mortality after adjusting for comorbidity Older patients have also been identified as having the lowest levels of NAD+ (Xie J.et al., 2015), while, conversely, those with the lowest risk, infants and children have the highest levels.

Oxidative stress also activates the NAD+-dependent enzyme, poly ADP ribose polymerase 1 (PARP1) (Yoo C.-Het al., 2014) hyperactivity of PARP1 results in depletion of cellular NAD+ pools, leading to ATP deficiency, energy loss, and subsequent cell death. These processes have the potential to enhance the pro-inflammatory cascade.

NAD+ deficiency impairs SIRT1 function (Guarente L et al., 2014) and its successful activation. Whereas extreme niacin deficiency is associated with the development of pellagra, more subtle decreases occur in diabetes, ageing PARP-1 is an abundant nuclear enzyme that modifies substrates by poly(ADP-ribose)-ylation. PARP-1 has well-described functions in DNA damage repair and also functions as a context-specific regulator of transcription factor

Oxidized and reduced Nicotinamide Adenine Dinucleotide (NAD+ and NADH respectively) are crucial metabolites in metabolic reactions. PARP-1 and PARP-2 use NAD+ as a cofactor in their catalytic activity. Continuous PARP activation can reduce intracellular levels of NAD+ by 80% and raises nicotinamide (NAM). SIRT1 is a NAD+-dependent protein deactelyase. (P. Bai et al., 2011) It has been known that the decrease of NAD+ and the increase of NAM ensured by enhanced PARP activity correlates with a downregulation of SIRT1 activity (J Biol Chem et al., 2005)similarly, the activation of SIRT1 reduced PARP activity. These observations raised four possible crosstalks between SIRT1, PARP-1

ELIGIBILITY:
Inclusion Criteria:

1. Patient adult age 18years and over(higher incidence) presented to Assiut University Hospital from 1december2020 to 30march.2021(winter2021-second wave)
2. Suspected of covid19 beacuse of the presence of symptoms suggestive of pneumonia (fever>38) and at least one of the following symptoms ;cough, dyspnea, tachpnea or hypoxia
3. having undergone RT-PCR (confirmed positive PCR)
4. Chest CT within 5 days of initial PCR

Exclusion Criteria:

1. Cases less than 18 years old
2. Cases express a dissent from the use of their data in the syudy
3. Cancer patients (affect result of study as they have disrubted level of these biomarker)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: COVID19 patient with clinical mainfastion with x.ray finding and positive PCR
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Sirtuin1 in COVID19 | 1 year
  The NAD dependent deacetylase activity of Sirtuin1 in COVID19

REFERENCES:
- [Background] Cardellini M, Menghini R, Martelli E, Casagrande V, Marino A, Rizza S, Porzio O, Mauriello A, Solini A, Ippoliti A, Lauro R, Folli F, Federici M. TIMP3 is reduced in atherosclerotic plaques from subjects with type 2 diabetes and increased by SirT1. Diabetes. 2009 Oct;58(10):2396-401. doi: 10.2337/db09-0280. Epub 2009 Jul 6. PMID 19581416
- [Background] Chung M, Bernheim A, Mei X, Zhang N, Huang M, Zeng X, Cui J, Xu W, Yang Y, Fayad ZA, Jacobi A, Li K, Li S, Shan H. CT Imaging Features of 2019 Novel Coronavirus (2019-nCoV). Radiology. 2020 Apr;295(1):202-207. doi: 10.1148/radiol.2020200230. Epub 2020 Feb 4. PMID 32017661
- [Background] Guarente L. Calorie restriction and sirtuins revisited. Genes Dev. 2013 Oct 1;27(19):2072-85. doi: 10.1101/gad.227439.113. PMID 24115767
- [Background] Siddiqi HK, Mehra MR. COVID-19 illness in native and immunosuppressed states: A clinical-therapeutic staging proposal. J Heart Lung Transplant. 2020 May;39(5):405-407. doi: 10.1016/j.healun.2020.03.012. Epub 2020 Mar 20. No abstract available. PMID 32362390